CLINICAL TRIAL: NCT00290459
Title: Prognostic Markers of Gynecologic Cancers
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Zhenmin Lei, Professor, University of Louisville
Other Study IDs: 608.03
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Gynecologic Disease; Gynecologic Cancer
Keywords: Gynecologic Disease; Gynecologic Cancer; Prognostic Markers
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other

SUMMARY:
This proposal seeks to retain "discard" pieces of human gynecologic tissues and "discard" ascites fluid collected during normal surgical procedures, along with corresponding blood samples and urine, for research involving prognostic markers of disease/cancer. The specific aims of the proposal include:

1. To collect "discard" pieces of benign, pre-malignant and malignant gynecologic tissues, "discard" ascites fluid and, when possible, corresponding blood and urine specimens from patients undergoing:

   1. hysterectomy
   2. excisions of cervical dysplasia and/or venereal warts, and
   3. therapeutic excisional surgeries to remove gynecologic disease/cancer (uterine, ovarian and lower female genital tract).
   4. paracentesis for the symptomatic relief of ascites fluid accumulation (distention).
2. To collect pre-operative blood and urine from patients along with pre- operative blood work drawn for clinical evaluation.
3. De-identify the patients from their donated tissue, blood and urine specimens by assigning a laboratory identification number.
4. Rapidly process and store the collected specimens to preserve biological integrity. (RNA, DNA and proteins)
5. Collect and record the patient's demographic and medical information into a research database under the assigned lab number only.
6. Assess the specimens for prognostic markers of gynecologic disease/cancer by molecular techniques such as DNA arrays,immunohistochemistry and ELISA.

DETAILED DESCRIPTION:
During the last two decades, cancer research has shifted from using cell lines and animal models to directly using human tissue. This is especially true for research focused on premalignancies for which there are few good animal models. Research utilizing human tissues and sera not only addresses many issues/questions of medical research that cannot be evaluated in cell lines and/or in animal models of human disease, but it also provides a system to test the relevance of these findings to human diseases. Various biologic and genetic changes that occur in the developmental stages of human neoplasia can be identified and analyzed using human tissues.

Research using human tissues and sera is making great strides in the effort to define possible markers of developing neoplasia and will promote the design of targeted cancer treatments and possible prevention. It is important to link research findings in tissue and blood specimens to the clinical outcome of patients with malignancy so we can pinpoint when and where, during the course of cancer development, molecular changes occur.

Many malignancies of the female genital tract may arise in more than one location, either synchronously or metachronously, giving rise to the concept of a "field" effect of carcinogenesis. By collecting tissue from multiple epithelial sites (sampled by the physician) it is possible to compare the molecular changes seen in preinvasive to those that occur in invasive neoplasia for differential expression profiles of potential markers. If protein markers are identified in cells present in the diseased tissue we can check the patient's serum and urine to see if the proteins can be detected. This information will enable us to screen and possibly identify these protein markers in patient serum and urine to correlate with the presence of a premalignant or malignant state.

Malignant ascites is excess fluid that accumulates in the space between the membranes lining the abdomen and abdominal organs, otherwise known as the peritoneal, or abdominal cavity. Malignant ascites typically occurs because of a disease, infection, or cancer in the peritoneal cavity that produces excessive fluid. Ascites fluid accumulation is very common in gynecologic cancers, especially ovarian. If protein markers are identified in the cells present in the diseased ascites fluid we may be able to correlate these markers with metastasis of the disease/cancer and possibly help prevent the spread of several gynecologic cancers.

ELIGIBILITY:
Inclusion Criteria:

* all female patients older than 18 years of age who are:
* undergoing hysterectomy
* excisions of cervical dysplasia and/or venereal warts
* therapeutic excisional surgeries for any benign or malignant gynecologic disease
* paracentesis procedure for the symptomatic relief of ascites fluid accumulation (distention)

Exclusion Criteria:

* women who are pregnant
* women who are HIV or Hepatitis C positive
* women who are enrolled in a current clinical trial utilizing the specimens

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female patients undergoing hysterectomy at the Brown Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 1321 (Actual)
Dates: Start 2003-12; Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhenmin Lei, MD, Principal Investigator — University of Louisville, James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- [Background] Chen Y, Miller C, Mosher R, Zhao X, Deeds J, Morrissey M, Bryant B, Yang D, Meyer R, Cronin F, Gostout BS, Smith-McCune K, Schlegel R., "Identification of Cervical Cancer Markers by cDNA and Tissue Microarrays," Cancer Research, Vol. 63(8), p.1927 - 1935, April 2003. Nucci MR, Castrillon DH, Bai H, Quade BJ, Ince TA, Genest DR, Lee KR, Mutter GL, Crum CP, "Biomarkers in Diagnostic Obstetric and Gynecologic Pathology: a Review," Adv. Anat. Pathol.,Vol.10(2), p. 55-68, March 2003. Nicolette CA, Miller GA., "The Identification of Clinically Relevant Markers and Therapeutic Targets," Drug Discov. Today, Vol. 8(1), p. 31-38, Jan. 2003. Salvesen HB, Akslen LA., "Molecular Pathogenesis and Prognostic Factors in Endometrial Carcinoma," APMIS, Vol. 110(10), p. 673-689, Oct. 2002. Geisler JP, Geisler HE, "Tumor Markers and Molecular Biological Markers in Gynecologic Malignancies," Curr. Opin. Obstet. Gynecol., Vol. 13(1), p. 31-39, Feb. 2001. Holschneider CH, Berek JS, "Ovarian Cancer: Epidemiology, Biology, and Prognostic Factors," Semin. Surg. Oncol., Vol. 19(1), p. 3-10, Jul-Aug 2000. Framarino dei Malatesta ML, Veneziano M, Peppicelli M, Lanzi G, Marzetti L, "Biologic Prognostic Factors in Ovarian Cancer: a Review," Eur. J. Gynaecol. Oncol., Vol. 19(2), p. 123-125, 1998. Busmanis I, "Biomarkers in Carcinoma of the Cervix: Emphasis on Tissue-Related Factors and their Potential Prognostic Factors," Ann. Acad. Med. Singapore, Vol. 27(5), p. 671-675, Sep. 1998. Grizzle WE, "Biomarkers - The New Frontier in the Pathology of Invasive and Preinvasive Neoplasias," Biotech. Histochem., Vol. 72(2), p. 59-61, March 1997. Grizzle WE, Myers RB, Manne U, "The Use of Biomarker Expression to Characterize Neoplastic Processes," Biotech. Histochem., Vol. 72(2), p. 96-104, March 1997.